CLINICAL TRIAL: NCT01194024
Title: Burn Multicenter Proposal: Development of an Inhalation Injury Scoring System to Predict Severity of Inhalation Injury
Brief Title: Scoring System for Inhalation Injury
Status: Completed | Type: Observational
Sponsor: American Burn Association (Other)
Collaborators: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: ABA-MCTG-0004
Record Dates: First submitted 2010-09-01; First posted 2010-09-02 (Estimated); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Inhalation Injury
Keywords: Inhalation Injury, Smoke; Inhalation Injury, Acute
MeSH Terms: conditions — Smoke Inhalation Injury | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — bronchioalveolar lavage specimens, blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Intubated within 24hrs of admission: All patients that are admitted to a participating burn center and intubated within 24 hours
  Interventions: Other: Standard of Care

INTERVENTIONS:
Other: Standard of Care — bronchoscopy with collection of bronchioalveolar lavage specimen, blood samples, High-Resolution spiral computed tomography(CT)

SUMMARY:
The goal of this multicenter study is to develop a standardized scoring system for inhalation injury that can be used both to quantify and predict injury severity inhalation injury in adults over 18 years of age. A model will be developed based on clinical, radiographic, bronchoscopic, and biochemical parameters that will predict the severity of inhalation injury with greater than 80% predictive accuracy

DETAILED DESCRIPTION:
The goal of this multicenter study is to develop a standardized scoring system for inhalation injury that can be used both to quantify and predict injury severity inhalation injury in adults over 18 years of age. A model will be developed based on clinical, radiographic, bronchoscopic, and biochemical parameters that will predict the severity of inhalation injury with greater than 80% predictive accuracy

ELIGIBILITY:
Inclusion Criteria:

* Injury consistent with inhalation of smoke or products of combustion
* Requires intubation within 24 hours of injury
* Meets one of the following 4 criteria

  1. history of closed space injury
  2. carbonaceous sputum
  3. elevated carboxyhemoglobin
  4. dx of inhalation injury is considered likely by investigator

Exclusion Criteria:

* ≤ 17 years of age
* Prisoner

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population includes all patients admitted to a participating burn center and who are intubated withing 24 hours of injury
  .
Sampling Method: Non-Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2011-11-30 (Actual); Primary Completion 2019-09-29 (Actual); Study Completion 2019-09-29 (Actual)

PRIMARY OUTCOMES:
Development of a diagnostic model to predict the severity of inhalation injury | within 48 hours of admission
  The development of a diagnostic model to predict the severity of inhalation injury based on demographics, characteristics of injury, bronchoscopy, CT scan, and inflammatory markers.

SECONDARY OUTCOMES:
Impact of inhalation injury | at discharge
  Assessment of the impact of inhalation injury on the incidence of pneumonia, acute respiratory distress syndrome (ARDS), and acute lung injury (ALI).

CONTACTS AND LOCATIONS:
Overall Officials: Kevin N. Foster, MD, Principal Investigator — The Arizona burn Center, Maricopa Integrated Health Systems
Locations (9):
- United States (9):
  - The Arizona Burn Center, Maricopa Integrated Health Systems, Phoenix, Arizona
  - Arkensas Children's Hopital, Little Rock, Arkansas
  - University of California Davis Medical Center, Sacramento, California
  - Loyola University, Maywood, Illinois
  - Indiana University, Indianapolis, Indiana
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - The Metro Health System, Cleveland, Ohio
  - University of Tennessee Health Science Center, Memphis, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas

REFERENCES:
- [Derived] Ronkar NC, Galet C, Richey K, Foster K, Wibbenmeyer L. Predictors and Impact of Pneumonia on Adverse Outcomes in Inhalation Injury Patients. J Burn Care Res. 2023 Nov 2;44(6):1289-1297. doi: 10.1093/jbcr/irad099. PMID 37352120